CLINICAL TRIAL: NCT03188016
Title: Feasibility Study: Improvised Music to Enhance the Effectiveness of Intensive Interaction in Developing Interpersonal Communication of Profoundly Intellectually Disabled Children and Young People
Brief Title: Improvised Music to Enhance Intensive Interaction Version 1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfavourable ethical opinion, principally on grounds of inadequate sample size
Sponsor: Beacon Hill Academy (Other)
Collaborators: The Music Therapy Charity Ltd (Unknown); Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Dr John B A Strange, Principal Investigator, Beacon Hill Academy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBASMT2; BHR/MT/SLT-1 (Other: Beacon Hill Academy)
Record Dates: First submitted 2017-06-10; First posted 2017-06-15 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Child Development Disorders, Specific; Developmental Communication Disorders
Keywords: "music therapy"; "Intensive Interaction"; "non-verbal communication"; "musical improvisation"; "feasibility study"; "randomised controlled trial"
MeSH Terms: conditions — Developmental Disabilities; Communication Disorders; Nonverbal Communication

STUDY DESIGN:
Intervention Model Description: Homogenous group randomly split into experimental and control groups to receive same number and duration of treatments
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are effectively masked since their parents/carers giving consent on their behalf will be masked regarding which arm their children are assigned to. (Participants themselves lack intellectual capacity to understand or consent to study participation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Interaction with music (Experimental): Weekly Intensive Interaction (Nind & Hewett) from a trained support worker plus music improvised by a music therapist with the aim of enhancing child - support worker interaction
  Interventions: Behavioral: Intensive Interaction with Music
- Standard Intensive Interaction (Active Comparator): Weekly Intensive Interaction (Nind & Hewett) from a trained support worker
  Interventions: Behavioral: Standard Intensive Interaction

INTERVENTIONS:
Behavioral: Intensive Interaction with Music — Intensive Interaction is a form of non-verbal communicative behaviour performed by a support worker to encourage and develop spontaneous communicative behaviour by the treatment subject, for which support workers are prepared by a speech and language therapist. The music in the intervention is live music improvised by a (UK) registered music therapist present in the room with treatment subject and support worker, who watches but does not participate socially in their interactions, and who develops musical input to encourage and enhance those interactions.
  Arms: Intensive Interaction with music
Behavioral: Standard Intensive Interaction — Intensive Interaction is a form of non-verbal communicative behaviour performed by a support worker to encourage and develop spontaneous communicative behaviour by the treatment subject, for which support workers are prepared by a speech and language therapist.
  Arms: Standard Intensive Interaction

SUMMARY:
The project will investigate the effectiveness of a specialised musical-clinical approach used as an adjunct to an established non-musical intervention in the enhancement of interpersonal interaction.

6 school pupils with profound disability will be randomly allocated to experimental and control groups. The control group will receive only Intensive Interaction for 16 sessions. The experimental group will receive four sessions of Intensive Interaction, followed by twelve sessions of Intensive Interaction plus improvised music. Music therapists will follow a flexible manual written to ensure that their music supports the interaction between pupil and learning support assistant (LSA) without direct social interaction with either.

Changes in capacity for interpersonal interaction will be assessed by a standardised assessment instrument, the Pre-Verbal Communication Schedule (PVCS), administered to both experimental and control groups before the 1st session and after the 16th session.

There will also be a qualitative process study of the experimental group conducted by video observation by the researchers involved.

The project is funded in equal shares by the Music Therapy Charity and Beacon Hill Academy.

DETAILED DESCRIPTION:
This is a small feasibility study to be conducted at a single research site, a special school for sensory and physical needs. The study is intended both to trial the research methodology and to estimate the effect size likely to be found if a larger study were carried out.

Intensive Interaction is a form of behavioural intervention developed by Nind and Hewett and extensively practised in schools and other institutions caring for people with profound intellectual disability who require special support in order to develop (non-verbal) interpersonal communication. Whilst the term Intensive Interaction can describe the attitude and behavioural style of staff throughout their contact with subjects, it can also, as in this study, refer to specific scheduled times in which the approach is adopted by staff with individual pupils or service users.

The subjects of this study are among those for whom Intensive Interaction is most beneficial, as assessed by the speech and language therapist at the research site. As these pupils would normally receive this intervention on account of their assessed needs, Intensive Interaction is designated the 'active comparator' (otherwise known as 'treatment as usual').

Since in the experimental condition two staff support each subject simultaneously, there is a need to distinguish effects attributable to the additional music from those attributable to the behaviour of the primary interactors. By treating Intensive Interaction as the active comparator it is hoped any effects of added music may be isolated.

Improvised music is in this study being trialed as an adjunctive therapy to Intensive Interaction. Previous research suggests that music improvised music therapist can under certain conditions facilitate the development of interpersonal interaction between subject and support worker. To replicate the conditions under which the previous study found this to be the case, the musical intervention has been manualised to guide the 2 music therapists who will provide the improvised supportive music. They will add music from session 5 of a total of 16, having observed the progress of Intensive Interaction without music during the first 4 sessions in order to make a detailed assessment of needs and how music might meet them.

A standardised assessment instrument, the Pre-Verbal Communication Schedule (PVCS), will be administered before each subject's first session of Intensive Interaction, and again after her/his 16th session to obtain a global view of non-verbal communicative behaviour. Pre- and post-test scores will be compared. The theoretical basis of both Intensive Interaction and the specific use of adjunctive improvised music is primarily affective, but it is important that any benefits should also be detectable in functional terms, hence the choice of PVCS rather than a more affectively orientated measure.

Additionally, qualitative data on the therapeutic process will be extracted from post-session notes and observations of video recordings of the sessions by those involved in the work with each participant.

Should the effectiveness of the specialised musical-clinical approach be supported by the results, a larger study could then establish the approach as an additional psycho-social resource for developing the interpersonal interaction skills of those with profound intellectual disability. The approach requires a modest level of additional training for a registered music therapist, but no additional qualification.

ELIGIBILITY:
Inclusion Criteria:

* the criteria the school normally applies, namely severely restricted capacity, and/or absent or limited motivation, for interpersonal interaction

Exclusion Criteria:

* any child who already receives Intensive Interaction or individual or small group music therapy or has done so in the previous school year.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-10-23 (Estimated); Primary Completion 2018-03-02 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Pre-Verbal Communication Schedule | 16 weeks between baseline measurement and outcome measurement
  A multi-element questionnaire administered face to face by a trained administrator to those most familiar with the subject (normally the parents/carers) to obtain a profile of communicative capacity and its application in all domains and an overall score. In this study those completing the questionnaire will be those staff most familiar with each participant (excluding those administering the experimental or control intervention.

CONTACTS AND LOCATIONS:
Overall Officials: John BA Strange, PhD, Principal Investigator — Voluntary research contract to Beacon Hill Academy
Locations (1):
- Beacon Hill Academy, South Ockendon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] http://davehewett.com/about-intensive-interaction
- [Background] Strange, J. (2017a) 'Assistants as Interaction Partners: The Experience of Learning Support Assistants in Group Music Therapy.' ' In J. Strange, H. Odell-Miller and E. Richards (eds) Collaboration and Assistance in Music Therapy Practice: Roles, Relationships, Challenges (pp. 22-35). London: Jessica Kingsley Publishers.
- [Background] Strange, J. (2017b) 'Improvised music to support client-assistant interaction: The perceptions of music therapists.' In J. Strange, H. Odell-Miller and E. Richards (eds) Collaboration and Assistance in Music Therapy Practice: Roles, Relationships, Challenges (pp. 235-252). London:Jessica Kingsley Publishers.
- Available data/document: PhD thesis explaining origin of the musical improvisation approach to be trialed — http://arro.anglia.ac.uk/314588/ — NB In the thesis the staff interacting with the young people with intellectual disability were not following principles of Intensive Interaction, although some had been trained in that approach and spontaneously applied some elements of it. All cases were studied solely by way of reviewing video recordings after a lapse of 1 - 2 years.